CLINICAL TRIAL: NCT05376774
Title: Prediction Model of Vitamin D Deficiency in Critically Ill Patients
Brief Title: Prediction Model of Vitamin D Deficiency
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202203073RIND
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness
Keywords: critical care; vitamin D
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Patients admitted to intensive care units
  Interventions: Other: Admitted to intensive care units

INTERVENTIONS:
Other: Admitted to intensive care units — Admitted to intensive care units

SUMMARY:
Many studies have pointed out that patients with vitamin D deficiency have a longer stay in the intensive care unit and a poor prognosis. Previous multi- center prospective observational study in Taiwan reveals that the prevalence of vitamin D deficiency in critically ill patients in northern Taiwan is 59%, and the prevalence of severe vitamin D deficiency is 18%. Several prediction models of vitamin D deficiency had been built for the general population but not patients admitted in intensive care units.

This multi-center retrospective study aims to develop and validate a score-based prediction model for severe vitamin D deficiency in critically ill patients. Investigators will review the data of previous multicenter, prospective, observational study. For temporal validation, the data will be divided into a derivation cohort (first 80% of the data set based on chronology) and a validation cohort (the remaining data set). The development and validation of the models will be carried out following the recommendations established in the Transparency Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD) initiative.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care units

Exclusion Criteria:

* aged < 20 years
* admitted to intensive care unit longer than 28 days
* body max index < 18 kg/m2
* receive vitamin D supplement > 3000 IU/day
* previously admitted to intensive care unit within 3 months
* have parathyroid disease, rickets, or severe liver cirrhosis [Child C]

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Performance of the score-based prediction model | 1 day
  Area under the receiver operating characteristic (AUROC) and area under precision recall curve (AUPRC) of the prediction models for severe vitamin D deficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No